CLINICAL TRIAL: NCT00894088
Title: A Single Dose, 2-Period, 2-Treatment 2-Way Crossover Bioequivalency Study of Mycophenolate Mofetil 500 mg Tablets Under Fasting Conditions
Brief Title: Bioequivalency Study of Mycophenolate Mofetil 500 mg Tablets Under Fasted Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Roxane Laboratories, Inc
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MYCO-T500-PVFS-1
Record Dates: First submitted 2009-05-04; First posted 2009-05-06 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Prophylaxis of Organ Rejection
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Mycophenolate Mofetil 500 mg Tablet
  Other Names: CellCept

SUMMARY:
The objective of this study was to prove the bioequivalence of Mycophenolate Mofetil 500 mg tablets under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C. Treatment with known enzyme altering drugs. History of allergic or adverse response to mycophenolate mofetil or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2006-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
bioequivalence determined by statistical comparison Cmax | baseline, 2-period, 14 day washout

CONTACTS AND LOCATIONS:
Overall Officials: William Allan Alexander, M.D., Principal Investigator — CEDRA Clinical Research
Locations (1):
- CEDRA Clinical Research, Austin, Texas, United States